CLINICAL TRIAL: NCT03361254
Title: Division and Cryopreservation of Autologous Blood Nuclear Cells for Intensive Regimen of Extracorporeal Photopheresis : Interest for the Treatment of Patients With Steroid Resistant Graft Versus Host Disease
Brief Title: Cryopreservation of White Blood Cells Before Their UVA Irradiation for Graft Versus Host Disease Treatment
Acronym: cryo-ECP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APJC2015/CRYOPCE-POCHON/NK
Record Dates: First submitted 2017-11-22; First posted 2017-12-04 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Graft Versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Cryopreservation

STUDY DESIGN:
Intervention Model Description: demonstrate the ability of this technique to follow high intensity regimen recommendations
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: cryopreservation — cryopreservation to every patient with an indication of ECP for acute or chronic GVHD in Nancy Hospital for 18 months

SUMMARY:
Extracorporeal photopheresis (ECP) is a worldwide recognized treatment of acute and chronic mild to moderate graft versus host disease (GVHD), in second or further line of treatment. Contrary to immunosuppressive drugs, ECP is not associated with side effects such as opportunistic infections, and is not associated with a higher frequency of relapse of the initial hematological disease. High intensity of ECP regimen (1 to 3 sessions per week, in case of chronic or acute GVHD) seems to be correlated to a higher efficacy. However, high intensity of ECP treatment is often difficult to sustain, because of frequent logistical problems to perform aphereses, such as venous access failure, infections of central line, deep blood cytopenias that require many transfusions before performing aphereses. Merlin et al. first described the feasibility of white blood cells cryopreservation before UVA irradiation, in vitro, then in vivo. We also recently reported the feasibility and efficacy of cryopreserved ECP in a series of 20 patients (adults and children), with acute and chronic GVHD, who had recurrent contraindications to aphereses, that prevented the realization of an intensive program of ECP. No adverse events occurred, and efficacy seemed to be similar to "classical" ECP (35% of complete overall response, and 40% of partial response). White blood cells (WBC) were divided after collection on Optia or Cellex apheresis machines: one was immediately treated with 8-MOP (methoxsalen) and ultraviolet A (UVA) irradiation, while the other was cryopreserved, and further (a few days later) thawed, sensitized with 8-MOP and irradiated before injection to the patient.

The aim of this study is to analyze this method in a prospective way, with complete biological data collection, of apoptosis, cytokines release etc…, necessary to the full description of cryopreservation of white blood cells before their irradiation and reinjection to the patient.

We will propose this technique of cryopreservation to every patient with an indication of ECP for acute or chronic GVHD in Nancy Hospital for 18 months.

DETAILED DESCRIPTION:
The main objective of this prospective interventional pilot study is to demonstrate the ability of this technique to follow high intensity regimen recommendations, as mentioned above:

* 3 ECP sessions (thawed or fresh) per week during 3 months for grade III to IV acute GVHD, then
* 2 ECP sessions (thawed or fresh) per week during 3 months for grade II acute GVHD
* 1 ECP session per week for chronic GVHD during 3 months

The other objectives are:

* To describe the safety and efficacy of cryo ECP. Efficacy will be assessed with a composite criteria test, comporting 5 items, which will be compared for each patient with a paired cohort of historical patients treated in Nancy University Hospital since 2010 (match will be made on type and grade of GVHD, and age under and over 18 year-old)
* To fully describe the biological consequences of cryopreservation of WBC before UVA irradiation: apoptosis rate and time, lymphocyte functional tests (lymphoblastic transformation test), cytokines release, number of lymphocytes, and monocytes at the time of reinjection, bacteriological tests, residual diméthylsulfoxyde (DMSO) quantification
* To demonstrate the decrease in red blood cells and platelets transfusion number, due to the sparing effect of cryo ECP on aphereses number.

ELIGIBILITY:
Inclusion Criteria:

* Adult or child who received an allogeneic hematopoietic stem cell transplantation, with a medical follow-up at the University Hospital of Nancy, or at the other University Hospitals in the great East region (Dijon, Reims, Besançon) in which ECP is not accessible.
* Eligible for ECP for the treatment of acute or chronic steroid refractory GVHD, after pluridisciplinary concertations
* Patients (or parents) who received full information on the research and who signed a consent for this research

Non inclusion Criteria:

* Children under 10 kg of weight
* Patients or parents who did not sign a consent
* Patients who present an absolute contra-indication for apheresis: recent pulmonary embolism, deep vein thrombosis, myocardial infarction, active and evolutive bacterial or fungal infection, hemodynamics instability, deep anemia (Hb < 8g/dl) or deep thrombocytopenia (< 20 g/L) despite transfusions, severe hypocalcemia.
* Women in age to procreate without contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2020-03-31 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
intensity of ECP regimen | 3 months after the first ECP session
  Number of ECP (fresh and thawed) sessions during 3 months

SECONDARY OUTCOMES:
systemic infections during 3 months after cryo-ECP (safety) | at 6 weeks and 3 months after the first ECP session
occurrence of death after cryo-ECP (safety) | at 6 weeks and 3 months after the first ECP session
occurrence of relapse of the initial hematological disease after cryo-ECP (safety) | at 6 weeks and 3 months after the first ECP session
Steroid sparing effect (efficacy) | at 6 weeks and 3 months after the first ECP session
GVHD grade (severity) (efficacy) | at 6 weeks and 3 months after the first ECP session
immunosuppressive drugs used (efficacy) | at 6 weeks and 3 months after the first ECP session